CLINICAL TRIAL: NCT05525182
Title: Efficacy and Safety of ES16001 in Patients With COVID-19: a Phase II/III, Multinational, Randomized, Parallel-group, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of ES16001 in Patients With COVID-19
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genencell Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GNC_ESE_COVID19_P2-301
Record Dates: First submitted 2022-07-21; First posted 2022-09-01 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Elaeocarpus sylvestris extract

STUDY DESIGN:
Intervention Model Description: Phase II -Dose-finding Phase II will be enrolled 424 patients (1:1:1:1 ratio) randomly assigned to one of the four treatment groups as follows.
  * ES16001 480 mg /day
  * ES16001 720 mg /day
  * ES16001 960 mg /day
  * Placebo
  Phase III In the phase III, safety and efficacy with the dose selected in the phase II will be compared with placebo. In the phase III, about 706 patients will be randomized in 1:1 ratio to test drug or placebo. Randomization will be stratified depending on the well-known risk factors for progression and disease severity of a patient. Final Endpoints and the sample size may be different depending on the results of the phase II.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, investigator staff and all site personnel will remain blinded to group allocation from randomization until database lock; randomization data will not be accessible by anyone involved in the study unless knowledge of the study treatment is relevant to the safety of the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase II (Experimental): ES16001: 480 mg/day ES16001: 720 mg/day ES16001: 960 mg/day Placebo
  Interventions: Drug: ES16001 40 mg; Drug: ES16001 80 mg; Drug: ES16001 160 mg; Drug: Placebo
- Phase III (Experimental): ES16001 Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ES16001 40 mg — Composition: Elaeocarpus extract 40mg tablet
  Other Names: 40 mg
  Arms: Phase II
Drug: ES16001 80 mg — Elaeocarpus extract 80 mg tablet
  Other Names: 80 mg
  Arms: Phase II
Drug: ES16001 160 mg — Elaeocarpus extract 160 mg tablet
  Other Names: 160 mg
  Arms: Phase II
Drug: Placebo — Placebo Tablet: Tablets for oral use indistinguishable from ES16001 in size, appearance, taste and smell

SUMMARY:
This is phase II/III, randomized, parallel-group, double-blind, placebo-controlled study. Patients must be at least 19 years of age (or according to the legal age for adult in each country) with confirmed mild or moderate COVID-19 tested positive with a real time reverse transcription polymerase chain reaction (RT-PCR) analysis of rhinopharynx samples. RT-PCR analysis of rhinopharynx samples must be <4 days old prior to the study enrolment

DETAILED DESCRIPTION:
After obtaining the consent and confirming eligibility, eligible patients will be treated with investigational medicinal product (IMP) for 7 days and followed up for additional 21 days (total 29 days). Patients who are discharged from the hospital or ending the quarantine may have to visit the investigational site on a pre-determined date for efficacy and safety follow up observation. Final safety and efficacy data will be collected on the last study day (29th Day).

If patients are fully recovered or discharged from the hospital prior to treatment period, all the evaluations on the 7th day/End of Treatment examination treatment shall be performed on the day of discharging.

ELIGIBILITY:
Inclusion Criteria:

1. Those with full understanding of the clinical study and agreeing with the participation of the clinical study voluntarily in writing, or with a deputy granted with legal authority of the relevant patient if he/she is unable to agree with the clinical study in person
2. Adults aged at 19 or above at the time of screening examination (according to the legal age for adult in each country)
3. Diagnosis of COVID-19 including a positive real time reverse transcription polymerase chain reaction (RT-PCR) for severe acute respiratory syndrome (SARS)-CoV-2 within 4 days prior to administering the investigational produce (IP)
4. mild or moderate patients who have the following conditions at screening and confirm at randomization at randomization A. Mild: Those with COVID-19 symptoms relevant to the inclusion criteria 5 without breathing difficulty or other chest radiation examination B. Moderate: Those with disease in respiratory organs in the clinical evaluation or imaging examination (chest radiation examination, etc.) and also relevant to the following conditions

   * Higher than 94% of oxygen saturation (Sp02) with room air at screening
   * Lower than 30 times/min respiratory frequency at screening
5. Those who happen more than one of the following symptoms within 4 days prior to the treatment of investigational medicinal product (IMP) and also have more than one of symptoms within a day prior to the treatment of IMP:

   * Fever
   * Cough
   * Shortness of breath
   * Chills
   * Muscle pain
   * Headache
   * Sore throat
   * Loss of smell/taste
   * Nasal congestion
   * Runny nose
   * Fatigue
   * Nausea or vomiting
   * Diarrhea
   * Phlegm
6. Those being hospitalized or scheduled in hospital or quarantined facilities or home isolated
7. Those comply with the clinical study protocol
8. Female patients of childbearing potential and male patients with partners of childbearing potential must agree to use adequate methods of contraception during the study and through 90 days after the last dose of study medication. Female patients of childbearing potential are all those except patients who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal. Effective contraception includes an established hormonal therapy or intrauterine device for females, and the use of a barrier contraceptive (i.e. diaphragm or condoms) with spermicide.

Exclusion Criteria:

1. Those with known or suspected hypersensitivity to ES16001 or any of its excipients
2. Those with genetic issues with galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption, etc.
3. Patients with ECG evidence of a QTcF > 450 ms in men and > 470 ms in women and patients with any other risk factors for Torsades de pointes (TdP) (hypokalemia, hypomagnesemia or hypocalcemia, family history of long QT syndrome, low left ventricular ejection fraction, left ventricular hypertrophy, ischemia and slow heart rate)
4. Concomitant use of hydroxychloroquine or other drugs known to prolong QT interval throughout the study 5. Suspected active bacterial, fungal, viral, or other infection (besides COVID-19).

6. Immunosuppressor or immunomodulatory drugs within the past 3 months (excluding corticosteroids) and patients with autoimmune disease.

7. Patients with one of the following severe COVID-19 signs at randomization (based on NIH classification)

* Oxygen saturation (SpO2) <94% of oxygen saturation without oxygen supply in room air
* Partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) <300 mmHg
* Respiratory frequency >30 times/min
* Parenchyma infiltration> 50% 8. Patients requiring oxygen treatment (nasal prong, facial mask, and high flow oxygen) or machine respiration (oxygen by NIV or high flow, intubation and mechanical ventilation, and etc.) at randomization 9. Those requiring extracorporeal membrane oxygenation (ECMO) or continuous renal replacement therapy (CRRT) treatment due to damage on multiple organs with severe illness (respiratory failure, shock, or multiple organ disorder) 10. Those with issues on kidney or liver as follows in the screening

  1. Alanine transaminase (ALT) or aspartate aminotransferase (AST) > 5 x upper limit of normal (ULN) at screening
  2. Total bilirubin that is 1.5 x upper limit of normal (ULN) at screening in the blood
  3. Serum creatine > 2mg/dL (> 176.8 μmol/L) or estimated creatine clearance < 30ml/min measured or calculated by Cockroft Gault equation 11. Absolute neutrophil count (ANC) <1000/μL in the screening 12. platelet count <50,000/μL in the screening 13. Those who are pregnant or breastfeeding 14. Treatment with an investigational product within 5 times half-life or to 30 days from the screening (whichever is longer) 15. Those taking antiviral drugs, anti-inflammatory medicine, or neutralizing antibody that is known to influence the treatment of COVID-19 (refer to 7.4.2 Prohibited medication) 16. Those with chronic disease that is inappropriate for the participation in clinical study judged by the investigator (Uncontrolled diabetes, chronic kidney disease, chronic liver disease, chronic lung disease, chronic cardiovascular disease, blood cancer, chemotherapeutic cancer patients, patients taking immunosuppressants, idiopathic thrombocytopenia, hyperkalemia patients, etc.)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase II | 2 months, last patient in (LPI) (Dec 22,23 respectively + 1 month Tx -> 2 months for database lock (DBL) and clinical study report (CSR)
  To determine the safe and effective dose of ES16001 versus placebo for the treatment of mild to moderate COVID-19. Proportion of subjects receiving the oxygen aiding treatment (nasal prong or facial mask) for at last 24 hours with oxygen saturation < 94% in room air prior to oxygen supply
  * Proportion of subjects requiring invasive machine ventilation as well as the non-invasive machine ventilation
  * Proportion of subjects applied with high flow oxygen or machine ventilation with oxygen saturation estimated to be less than 94% in room air
  * Proportion of dead subjects
Phase III | 2 months, last patient in (LPI) (Dec 22,23 respectively + 1 month Tx -> 2 months for database lock (DBL) and clinical study report (CSR)
  To demonstrate the superiority of ES16001 versus placebo for the treatment of mild to moderate COVID-19. Proportion of subjects receiving the oxygen aiding treatment (nasal prong or facial mask) for at last 24 hours with oxygen saturation < 94% in room air prior to oxygen supply
  * Proportion of subjects requiring invasive machine ventilation as well as the non-invasive machine ventilation
  * Proportion of subjects applied with high flow oxygen or machine ventilation with oxygen saturation estimated to be less than 94% in room air
  * Proportion of dead subjects

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyun Park, Study Chair — Genencell
Locations (3):
- South Korea (3):
  - Soon Chun Hyang University Hospital, Bucheon-si
  - Eunpyeong, St.Mary's Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No